CLINICAL TRIAL: NCT03124199
Title: Rifaximin Associated With Classic Triple Therapy (Inhibitor of Proton Pump, Amoxicillin and Clarithromycin) for the Eradication of Helicobacter Pylori Infection
Brief Title: Rifaximin Associated With Classic Triple Therapy for the Eradication of Helicobacter Pylori Infection
Acronym: R+OCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R+OCA
Record Dates: First submitted 2016-04-07; First posted 2017-04-21 (Actual); Results first posted 2018-02-19 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori)
Keywords: Eradication; Helicobacter pylori; rifaximin; therapy; standard triple therapy
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifaximin (Experimental): Patient with Helicobacter pylori infection with standard triple therapy prescribed by clinical practice.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 400 mg/8 h added to the standard triple therapy

SUMMARY:
Background: A progressive decrease in Helicobacter pylori eradication rates has been described over the years, so new combinations of antibiotics for treatment are needed.

Aim: To evaluate the efficacy and safety of the addition of rifaximin to standard triple therapy (omeprazole, amoxicillin and clarithromycin) for the eradication of H. pylori.

Methods: Independent prospective pilot clinical trial (EUDRA CT: 2013-001080-23). Forty consecutive adult patients were included with H. pylori infection, dyspeptic symptoms and naive to eradication treatment. A full blood test was performed in the first 5 patients included to evaluate the safety of the treatment. H. pylori eradication was confirmed with urea breath test at least 4 weeks after the end of treatment. Treatment: Rifaximin 400 mg/8 h, clarithromycin 500 mg/12 h, amoxicillin 1 g/12 h, and omeprazole 20 mg/12 h for 10 days.

DETAILED DESCRIPTION:
4. STUDY DESIGN 4.1. Endpoints Main endpoint Eradication of infection "by intention to treat". Secondary endpoints Eradication of infection "per protocol". Adherence to treatment. Medication side effects.

Clinical and demographic variables:

1) Age; 2) Sex; 3) Smoking habit; 4) Comorbidity (diabetes mellitus, hypertension, ischemic heart disease, dyslipidemia, others); 5) Indication of eradication (peptic ulcer vs. functional dyspepsia or not investigated) 6) Initial diagnosis test of H. pylori infection.

4.2. Clinical trial design Phase III clinical trial, prospective, pilot, open, not controlled. The recruitment period will be five months. All the tests to confirm infection with Helicobacter pylori made within a maximum period of one year, provided the patient has not taken any antibiotics able to eradicate bacteria from conducting the test until the day of inclusion, will be given as valid, for the inclusion of the patient, Patients with proven infection and that have already prescribed standard triple therapy by routine clinical practice, will be required written informed consent to participate in the study, after which treatment with Rifaximin will be added.

1. At the time of enrollment, after reviewing the inclusion and exclusion criteria and obtaining the patient's consent, a medical history and complete examination will take place including: antiulcer treatment received, history of smoking and alcohol intake, aspirin consumption and NSAID. Other concomitant medications that the patient is receiving for any other process will be also recorded.
2. Between days 5-15 after taking the last dose, the procedures of the follow up visit specified in section 7.3.2 will be performed to the patients. Similarly, these procedures will be performed at the time when the patient leaves the study prematurely, if need be.
3. Control breath test or histology between 4 and 8 weeks after treatment ends. Before the control test, it will be confirmed that the patient has not taken proton pump inhibitors during the 15 days before or antibiotics within 4 weeks prior to the breath test.

The breath test is approved for the detection of H. pylori infection and post-eradication control. Sample collection can be performed in the same hospital.

Breath test has been chosen as post-eradication control because it is the test that, in isolation, has a higher diagnostic accuracy, so is currently considered as the diagnostic method of choice to confirm eradication of H. pylori. In cases of gastric ulcer where gastroscopy after treatment control is required, the biopsy is valid also as post-eradication control.

A single test post-treatment control is requested at least four weeks after completion of therapy since it has been observed an excellent correlation between it and the long-term results in previous studies.

4.3. Treatment Description Control treatment: N/A Experimental treatment: rifaximin 400 mg (2 tablets of Rifaximin 200 mg)/8 hours for 10 days.

Study medication will be donated by "Alfa Wassermann" and re-labeled in accordance with the recommendations of the Royal Decree 223/2004 for medication trials.

4.5. Withdrawal criteria and analysis The patient can discontinue his/her participation in the study at any time he/she wishes. In his opinion and judgment, the researcher doctor may also decide to withdraw a patient from the trial if it does not comply with the protocol.

The occurrence of chronic diseases during the trail will result in the permanent exclusion of the subject. The onset of acute pathology during the trial period will delay the administration of test drugs until the patient is healed. Patients who may vomit within 3 hours after taking the drug (verified by asking the patient) or other clinically relevant process that may affect the pharmacokinetics of study drug, will be excluded from analysis Only subjects excluded from the trial before receiving the study medication will be replaced by others, so that the number of patients will remain as provided by the sample size calculation. Individual sheets of collecting data from these excluded subjects will also be sent to the Sponsor organization for evaluation.

4.6. Investigational drug accountability procedures Patients will receive Rifaximin and will be asked to return the remaining investigational medication in follow up visit after treatment. They will be asked to collaborate also bringing the remains of standard triple therapy for counting. The doctor will ask the patient about treatment compliance and count the residual medication after which he will return the remains of the standard triple therapy to the patient and preserve the remains of Rifaximin for later destruction by appropriate methods.

4.8. Definition of end of trial Date on which the last patient completed the study follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Patients with dyspeptic symptoms, ie pain or discomfort (including abdominal bloating, early satiety and bloating) centered on the upper abdomen, persistent or recurrent, with proven H. pylori infection (through testing breath or gastric biopsy based methods, if it has been done) with a validity period of one year.
3. Having been previously prescribed by routine clinical practice the standard triple therapy as eradication treatment:

   * Proton Pump Inhibitor. Omeprazole 40 mg (or equivalent) every 12 hours. Treatment duration: 10 days.
   * Clarithromycin. Dose: 500 mg every 12 hours. Treatment duration: 10 days.
   * Amoxicillin. Dose: 1000 mg every 12 hours. Treatment duration: 10 days.
4. Not having yet begun taking the eradication therapy.
5. Written informed consent from the patient.
6. The first five patients included in the study, should had cited from the outpatient and prior to his arrival in consultation, a routine analysis in the month after the completion of the eradication therapy.
7. If the patient is a woman of childbearing age, she will be asked to commit to not get pregnant or to use an adequate contraception method.

Exclusion Criteria:

1. Previous eradication treatment for H. pylori (these patients are often carriers of antibiotic resistant strains and have a much lower response than those that had never received treatment).
2. Allergy to any of the antibiotic in the treatment.
3. Taking antibiotics or bismuth salts since performing the breath test.
4. Previous gastric surgery.
5. Presence of severe pulmonary, hepatic, renal, endocrine, metabolic, hematologic or tumor disease.
6. Very advanced chronic disease or other conditions that prevent attending to controls and follow ups.
7. Previous history of alcohol or drugs abuse.
8. Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Perez, Gisbert, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gisbert JP, Calvet X, Bermejo F, Boixeda D, Bory F, Bujanda L, Castro-Fernandez M, Dominguez-Munoz E, Elizalde JI, Forne M, Gene E, Gomollon F, Lanas A, Martin de Argila C, McNicholl AG, Mearin F, Molina-Infante J, Montoro M, Pajares JM, Perez-Aisa A, Perez-Trallero E, Sanchez-Delgado J. [III Spanish Consensus Conference on Helicobacter pylori infection]. Gastroenterol Hepatol. 2013 May;36(5):340-74. doi: 10.1016/j.gastrohep.2013.01.011. Epub 2013 Apr 18. No abstract available. Spanish. PMID 23601856
- [Background] Gisbert JP, Pajares R, Pajares JM. Evolution of Helicobacter pylori therapy from a meta-analytical perspective. Helicobacter. 2007 Nov;12 Suppl 2:50-8. doi: 10.1111/j.1523-5378.2007.00576.x. PMID 17991177
- [Background] Graham DY. Helicobacter pylori eradication therapy research: Ethical issues and description of results. Clin Gastroenterol Hepatol. 2010 Dec;8(12):1032-6. doi: 10.1016/j.cgh.2010.07.002. Epub 2010 Jul 23. PMID 20656062
- [Background] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Background] Hawkey CJ, Atherton JC, Treichel HC, Thjodleifsson B, Ravic M. Safety and efficacy of 7-day rabeprazole- and omeprazole-based triple therapy regimens for the eradication of Helicobacter pylori in patients with documented peptic ulcer disease. Aliment Pharmacol Ther. 2003 Apr;17(8):1065-74. doi: 10.1046/j.1365-2036.2003.01492.x. PMID 12694089
- [Background] Paoluzi P, Iacopini F, Crispino P, Nardi F, Bella A, Rivera M, Rossi P, Gurnari M, Caracciolo F, Zippi M, Pica R. 2-week triple therapy for Helicobacter pylori infection is better than 1-week in clinical practice: a large prospective single-center randomized study. Helicobacter. 2006 Dec;11(6):562-8. doi: 10.1111/j.1523-5378.2006.00459.x. PMID 17083378
- [Background] Veldhuyzen Van Zanten S, Machado S, Lee J. One-week triple therapy with esomeprazole, clarithromycin and metronidazole provides effective eradication of Helicobacter pylori infection. Aliment Pharmacol Ther. 2003 Jun 1;17(11):1381-7. doi: 10.1046/j.1365-2036.2003.01554.x. PMID 12786632
- [Background] Vakil N, Lanza F, Schwartz H, Barth J. Seven-day therapy for Helicobacter pylori in the United States. Aliment Pharmacol Ther. 2004 Jul 1;20(1):99-107. doi: 10.1111/j.1365-2036.2004.02029.x. PMID 15225176
- [Background] Laine L, Fennerty MB, Osato M, Sugg J, Suchower L, Probst P, Levine JG. Esomeprazole-based Helicobacter pylori eradication therapy and the effect of antibiotic resistance: results of three US multicenter, double-blind trials. Am J Gastroenterol. 2000 Dec;95(12):3393-8. doi: 10.1111/j.1572-0241.2000.03349.x. PMID 11151867
- [Background] Laine L, Suchower L, Frantz J, Connors A, Neil G. Twice-daily, 10-day triple therapy with omeprazole, amoxicillin, and clarithromycin for Helicobacter pylori eradication in duodenal ulcer disease: results of three multicenter, double-blind, United States trials. Am J Gastroenterol. 1998 Nov;93(11):2106-12. doi: 10.1111/j.1572-0241.1998.00602.x. PMID 9820381
- [Background] Calvet X, Ducons J, Bujanda L, Bory F, Montserrat A, Gisbert JP; Hp Study Group of the Asociacion Espanola de Gastroenterologia. Seven versus ten days of rabeprazole triple therapy for Helicobacter pylori eradication: a multicenter randomized trial. Am J Gastroenterol. 2005 Aug;100(8):1696-701. doi: 10.1111/j.1572-0241.2005.50019.x. PMID 16086704
- [Background] Gisbert JP, Dominguez-Munoz A, Dominguez-Martin A, Gisbert JL, Marcos S. Esomeprazole-based therapy in Helicobacter pylori eradication: any effect by increasing the dose of esomeprazole or prolonging the treatment? Am J Gastroenterol. 2005 Sep;100(9):1935-40. doi: 10.1111/j.1572-0241.2005.00178.x. PMID 16128936
- [Background] Della Monica P, Lavagna A, Masoero G, Lombardo L, Crocella L, Pera A. Effectiveness of Helicobacter pylori eradication treatments in a primary care setting in Italy. Aliment Pharmacol Ther. 2002 Jul;16(7):1269-75. doi: 10.1046/j.1365-2036.2002.01244.x. PMID 12144576
- [Background] Altintas E, Sezgin O, Ulu O, Aydin O, Camdeviren H. Maastricht II treatment scheme and efficacy of different proton pump inhibitors in eradicating Helicobacter pylori. World J Gastroenterol. 2004 Jun 1;10(11):1656-8. doi: 10.3748/wjg.v10.i11.1656. PMID 15162544
- [Background] Gumurdulu Y, Serin E, Ozer B, Kayaselcuk F, Ozsahin K, Cosar AM, Gursoy M, Gur G, Yilmaz U, Boyacioglu S. Low eradication rate of Helicobacter pylori with triple 7-14 days and quadriple therapy in Turkey. World J Gastroenterol. 2004 Mar 1;10(5):668-71. doi: 10.3748/wjg.v10.i5.668. PMID 14991935
- [Background] Howden CW, Hunt RH. Guidelines for the management of Helicobacter pylori infection. Ad Hoc Committee on Practice Parameters of the American College of Gastroenterology. Am J Gastroenterol. 1998 Dec;93(12):2330-8. doi: 10.1111/j.1572-0241.1998.00684.x. No abstract available. PMID 9860388
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Egan BJ, Marzio L, O'Connor H, O'Morain C. Treatment of Helicobacter pylori infection. Helicobacter. 2008 Oct;13 Suppl 1:35-40. doi: 10.1111/j.1523-5378.2008.00639.x. PMID 18783520
- [Background] Yakoob J, Abid S, Abbas Z, Jafri SN. Antibiotic susceptibility patterns of Helicobacter pylori and triple therapy in a high-prevalence area. Br J Biomed Sci. 2010;67(4):197-201. doi: 10.1080/09674845.2010.11730319. PMID 21294447
- [Background] Vakil N, Hahn B, McSorley D. Clarithromycin-resistant Helicobacter pylori in patients with duodenal ulcer in the United States. Am J Gastroenterol. 1998 Sep;93(9):1432-5. doi: 10.1111/j.1572-0241.1998.455_t.x. PMID 9732920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty consecutive adult patients were included with H. pylori infection, dyspeptic symptoms and naive to eradication treatment
Pre-assignment Details: There were no significant events in the study after patient enrollment and before assignment
Period: Overall Study
Arm/Group | Rifaximin
Started | 40
Completed | 36
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Rifaximin
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Region of Enrollment [Number; unit: participants]
  Spain | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With H.Pylori Infection Eradication
Description: Percentage of Participants with H.Pylori Infection Eradication confirmed with urea breath test at least 4 weeks after the end of treatment
Time Frame: 1 month
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rifaximin
Number analyzed (Participants) | 40
percentage of participants | 61 [45 to 77]

2. Secondary Outcome: Tolerability of Treatment
Description: Patients with side effects present during treatment and in the 4 weeks after end of treatment
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Rifaximin
Number analyzed (Participants) | 36
participants
  with diarrhea | 13
  with metallic taste | 9
  headache | 5
  nausea | 5
  abdominal pain | 1

3. Secondary Outcome: Compliance With Treatment of Patients That Completed the Study
Description: Percentage of patients that has comply with treatment, considered as intake of more than 90% of study drugs in patients who attended the post-treatment visit.
Time Frame: 1 month
Measure: Number; unit: percentage of participants
Arm/Group | Rifaximin
Number analyzed (Participants) | 36
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: 1 month and 10 days
Arm/Group | Rifaximin
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 27/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin (N=36)
Diarrhea (Gastrointestinal disorders) | 13 — Diarrhea
Metallic Taste (Gastrointestinal disorders) | 9 — Metallic Taste
Headache (General disorders) | 5 — Headache
Nausea (Gastrointestinal disorders) | 5 — Nausea
abdominal pain (Gastrointestinal disorders) | 1 — Abdominal pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No